CLINICAL TRIAL: NCT04059796
Title: Clinical Investigation of OMEGA Gemini Capsule, Model Gemini Capsule 3 Rev 2 in Combination With a Commercially Available, FDA Approved Monofocal or Toric Intraocular Lens
Brief Title: Comparison of Gemini III Rev 2 Implanted in Conjunction With an Approved IOL vs Eyes Implanted With an Approved IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omega Ophthalmics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gemini III Rev 2
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be masked to which eye receives the study device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Eye (Experimental): Study device in conjunction with an approved monofocal or toric IOL after cataract extraction
  Interventions: Device: Omega Gemini III Rev 2 Device
- Control Eye (Active Comparator): approved monofocal or toric IOL after cataract extraction
  Interventions: Device: Control Eye

INTERVENTIONS:
Device: Omega Gemini III Rev 2 Device — Eyes randomized to receive the Gemini III Rev 2 device will receive the study device in conjunction with an approved monofocal or toric IOL post cataract extraction
  Arms: Study Eye
Device: Control Eye — Control eyes will receive an approved monofocal or toric IOL post cataract extraction
  Arms: Control Eye

SUMMARY:
This study is a prospective, observational, randomized, controlled, paired eye, subject-masked design.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to which eye will receive the Omega capsule Gemini 3 with an approved monofocal or Toric intraocular lens. Fellow eyes will receive an approved monofocal or Toric IOL (no Omega capsule).

Eyes randomized to receive one of the Gemini capsules (both models) will be eligible to have a secondary procedure (post 1-month postoperative visit) to correct refractive error.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older at the time of surgery diagnosed with bilateral cataracts
* Able to understand and sign an informed consent
* Willing and able to complete all study visits and assessments required for the study
* Calculated lens power within the available range
* Corrected distance visual acuity is equal to or worse than 20/40 in each eye with or without a glare source present
* Bilateral cataracts eligible for extraction by phacoemulsification and capsular bag fixated IOL implantation
* Potential postop visual acuity of 20/25 or better in the judgment of the surgeon
* Preoperative corneal astigmatism of 4.0 D or less with normal corneal topography
* Clear intraocular media other than cataract
* Preop endothelial cell density of 2000 cells/mm2 or more

Exclusion Criteria:

* Subject's best corrected vision is light perception or no light perception in either eye
* Cataract opacification preventing adequate Binocular Indirect Ophthalmoscopic retinal and macular examination.
* Orbital abnormalities, such as thyroid related orbitopathy, causing significant exophthalmos.
* Eyelid abnormalities causing lagophthalmos.
* Significant anterior blepharitis or meibomian gland dysfunction
* Corneal abnormalities or conditions, other than regular topographic corneal astigmatism
* Krukenburg's spindle (linear pigmentary deposits on the corneal endothelium)
* Abnormalities of the iris including trans-illumination defects
* Pupil abnormalities (abnormally shaped, fixed or non-reactive)
* Pharmacologic dilation less than 7 mm
* Axial length <22.5mm
* Lens thickness <4.1 mm
* Anterior chamber depth >2.8mm
* Extremely shallow anterior chamber <2.0mm
* Prior ocular surgery
* Epiretinal membrane
* Macular edema
* Retinal tears including operculated holes
* Amblyopia
* Glaucoma of any kind
* Pseudoexfoliation syndrome
* History of uveitis/iritis
* Diabetic retinopathy
* Acute, chronic or uncontrolled systemic or ocular disease that may confound the results of the study (including rheumatologic conditions such as Rheumatoid arthritis, ankylosing spondyliltis, Sjögren's syndrome, and neurologic conditions such as optic neuritis or multiple sclerosis).
* Prior or anticipated use of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) or similar medications
* Average Keratometry <38D or > 48D by topography
* Any pathology of the zonules including evidence of zonular weakness, zonular instability, zonular damage, or coloboma effecting zonules.
* History of ocular trauma
* Pregnant, lactating, or has another condition with associated fluctuation of hormones that could lead to refractive changes

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Absence of fusion of peripheral anterior and posterior capsule to the intraocular lens | 6 month Postop Visit
  Via dilated slit lamp examination subjects will be assessed for anterior and posterior Via dilated slit lamp examination subjects will be assessed for anterior and posterior fusion of the IOL to the capsular bag with a dichotomous "Yes/No" response.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Orlich, MD, Principal Investigator
Locations (1):
- Clinica 20/20, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No